CLINICAL TRIAL: NCT04193163
Title: Prospective Observational Clinical Study Conducted Over a 10-year Period on Patients Who Received the ESOP 2 Stem to Restore Joint Function, in Order to Confirm Security and Performance of the Device
Brief Title: Observational Study Conducted on Patients Receiving the ESOP 2 Stem to Confirm Security and Performance of the Device
Acronym: ESOP2
Status: Terminated | Type: Observational
Why Stopped: Discontinuation of the studied medical device on the market and not enough inclusion in the study.
Sponsor: FH ORTHO (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018-37
Record Dates: First submitted 2019-11-28; First posted 2019-12-10 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Hip Disease; Hip Fractures
Keywords: Arthroplasty; Hip replacement
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients receiving ESOP 2 stem
  Interventions: Device: Hip prosthesis - ESOP 2 cementless femoral stem

INTERVENTIONS:
Device: Hip prosthesis - ESOP 2 cementless femoral stem — ESOP 2 femoral stems are intended to be implanted in the femoral region during total hip arthroplasty in order to restore joint function.

SUMMARY:
This study is a post-market clinical follow-up conducted in order to collect long-term data on security and performance of the ESOP 2 stem, which is intended to be implanted in case of total hip replacement, when used in real life conditions according to the instructions for use.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the security of the ESOP 2 stem by calculating the survival rate up to 10 years of follow-up.

The secondary objectives are to evaluate the security and performance of the device by assessing radiological data, gathering complications and evaluating functional score and quality of life score up to 10 years of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Subject implanted with ESOP 2 stem in one of the following indication according to the instructions for use: hip disorders; femoral neck fracture
* Subject who received an information form and is willing to participate in the study

Exclusion Criteria:

* Contraindications described in the instructions for use
* Usual surgical contraindications
* Subject who is not able to express his/her non-opposition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from participating hospitals will be enrolled as part of their clinical routine care.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Survival rate | 10 years post-op

SECONDARY OUTCOMES:
Radiographies evaluation | immediate post-op, 3 months post-op, 1 year post-op, 5 years post-op, 10 years post-op
  Radiological results such as stability, osteointegration will be evaluated.
Rate of complications | per-op, 3 months post-op, 1 year post-op, 5 years post-op, 10 years post-op
  All complications will be gathered during intervention and up to 10 years postoperatively.
Functional outcomes such as pain, mobility | pre-op, 3 months post-op, 1 year post-op, 5 years post-op, 10 years post-op
  Functional outcomes will be determined by the Harris Hip score. This score ranges from 0 to 100, where, the higher the score, the better the patient outcome.
Quality of life evaluation | pre-op, 3 months post-op, 1 year post-op, 5 years post-op, 10 years post-op
  Quality of life will be determined by the OXFORD-12 score. This score ranges from 12 points to 60 points, where, the higher the score, the better the patient outcome.

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Clinique Tivoli Ducos, Bordeaux
  - Nouvelle Clinique Bel-Air, Bordeaux
  - CH Pasteur, Colmar
  - Clinique du Val d'Ouest, Écully
  - CH Raymond POINCARE, Garches
  - CH de Haguenau, Haguenau
  - Groupe Hospitalier Pitié-Salpêtrière, Paris

IPD SHARING:
Plan to Share IPD: No